CLINICAL TRIAL: NCT04136054
Title: Better Sleep in Psychiatric Care - Depression, Anxiety and PTSD. A Randomized Naturalistic Study of a Psychological Group Treatment for Sleep Problems in Psychiatric Patients With Depression, Anxiety and PTSD.
Brief Title: Better Sleep in Psychiatric Care - Depression, Anxiety and PTSD
Acronym: BSIP-DAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Susanna Jernelöv, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/80-31/1.1
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Sleep Problem; Anxiety Disorders; Affective Disorder
Keywords: Cognitive Behaviour Therapy; Psychological Intervention
MeSH Terms: conditions — Parasomnias; Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjusted group CBT-i for Depression, Anxiety and PTSD (Experimental): Cognitive Behavioral group intervention for sleep problems in patients with Depression, Anxiety and PTSD, based on Cognitive Behavioral Therapy for insomnia
  Interventions: Behavioral: Adjusted group CBT-i for Depression, Anxiety and PTSD
- Care as usual wait-list control group (Active Comparator): Treatment as Usual. (After about five months, participants in this condition are offered the experimental group treatment.)
  Interventions: Other: Care as usual wait-list control group

INTERVENTIONS:
Behavioral: Adjusted group CBT-i for Depression, Anxiety and PTSD — Adjusted group CBT-i for Depression, Anxiety and PTSD. CBT-i includes sleep scheduling/sleep compression, stimulus control, relaxation, cognitive interventions and sleep hygiene advice. Adjustments include the relationship between sleep and the psychiatric conditions at hand and and working with motivational enhancement techniques to increase adherence to treatment.
  Arms: Adjusted group CBT-i for Depression, Anxiety and PTSD
Other: Care as usual wait-list control group — Usual care at the clinic. This entails managing pharmacological treatment for the psychiatric problems and/or sleep problems. The clinic also provides different group treatments, such as mindfulness groups and CBT groups for symptoms of worry and depression, and individual therapy.
  Arms: Care as usual wait-list control group

SUMMARY:
Cognitive Behavioral Therapy (CBT) is treatment of choice for insomnia. Many patients in psychiatric care have sleep problems including insomnia, but are rarely given the choice to participate in CBT to improve their sleep. Patients with PTSD, Anxiety disorders and Depression display high levels of sleep difficulties. Sleep problems are often general, such as insomnia and sleep phase problems. In a previous pilot study, the investigators of the current study developed a CBT protocol that would target sleep problems in this mixed psychiatric population. The basis was CBT for insomnia (CBT-i), but also including techniques that would alleviate sleep phase problems (e.g. the systematic use of light and darkness), and techniques to target more general sleep related problems (e.g. difficulties waking up in the morning), that are also common in psychiatric patients. This treatment was well tolerated and gave large withing-group effects on insomnia severity in the pilot study. In a naturalistic randomized controlled trial, the investigators now evaluate the effects of this psychological treatment on sleep and anxiety and depressive symptoms in patients at the units for Anxiety and Affective disorders and Trauma, Southwest Psychiatry and Northern Stockholm Psychiatry, Stockholm County Council, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient at the clinics involved in the project
* Experiencing sleep problems (subjective report)
* Being able to participate in a psychological intervention in group format

Exclusion Criteria:

* Night shift work

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Changes from base-line to 8 weeks, 5 months and 14 months
  7-item, self-rated questionnaire measuring insomnia severity. Total score 0-28, higher score indicates more severe sleep problems.

SECONDARY OUTCOMES:
Actigraphy | Changes from base-line to post 8 weeks
  An actigraph is placed on the participant's arm for one week. It measures participants' arm-movements. An algorithm can be used to estimate sleep from movement data.
WHO Disability Assessment Schedule (WHODAS) | Changes from base-line to 8 weeks, 5 months and 14 months
  12-items self-rating questionnaire measuring disability. Total score (0-48), with higher score indicating more severe disability.
Patient Health Questionnaire (PHQ-9) | Changes from base-line to 8 weeks, 5 months and 14 months
  9-items self-rating questionnaire measuring level of depression. Total score 0-27 with higher score indicating more severe depression
Generalized Anxiety Disorder 7-item scale (GAD-7) | Changes from base-line to 8 weeks, 5 months and 14 months
  7-item self-rating questionnaire measuring level of anxiety. Total score 0-21 with higher score indicating more severe anxiety.
Sleep habits and behaviors | Changes from base-line to 8 weeks, 5 months and 14 months
  Self-rating questionnaire regarding the use of sleep promoting behaviors. The questionnaire was constructed for the larger BSIP project and consists of two parts. The first part includes statements such as "Last week I got out of bed within 15 minutes of waking up" to be answered by number of days the last week this was true (i.e. from 0 to 7). The second part is to be answered on a 6-point Likert scale from "Not at all true" to "Entirely true", with 7 statements like "I get out of bed the same time every morning". No total score is obtained.
Daytime Insomnia Symptoms | Changes from base-line to 8 weeks, 5 months and 14 months
  7-item self-rating questionnaire regarding daytime symptoms commonly associated with sleep problems. Total score 0-70, with higher score indicating more severe daytime symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Jernelöv, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Program for Affective disorders, Anxiety and Trauma, Stockholm Southwest Psychiatry, Stockholm, Sweden

REFERENCES:
- [Background] Cassel M, Blom K, Gatzacis J, Renblad P, Kaldo V, Jernelov S. Clinical feasibility of cognitive behavioural therapy for insomnia in a real-world mixed sample at a specialized psychiatric outpatient clinic. BMC Psychiatry. 2022 Sep 9;22(1):600. doi: 10.1186/s12888-022-04231-4. PMID 36085009